CLINICAL TRIAL: NCT05596435
Title: Early Detection of Pancreatic Cancer Using Plasma Cell-free DNA Fragmentomics
Brief Title: Early Detection of Pancreatic Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PANC-2022
Record Dates: First submitted 2022-10-24; First posted 2022-10-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma Cell-free DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Stage I-III pancreatic cancer: Cell-free DNA collected from plasma samples of 260 patients with stage I-III pancreatic cancer will undergo whole-genome sequencing
  Interventions: Other: No intervention
- Pancreatic disease: Cell-free DNA collected from plasma samples of 80 patients with pancreatic benign disease will undergo whole-genome sequencing
  Interventions: Other: No intervention
- Healthy controls: Cell-free DNA collected from plasma samples of 100 non-cancer individuals will serve as controls
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The purpose of this study is to enable non-invasive early detection of pancreatic cancer in high-risk populations through the establishment of a machine learning model using plasma cell-free DNA fragmentomics. Plasma cell-free DNA from early stage pancreatic cancer patients and healthy individuals will be subjected to whole-genome sequencing. Features, such as cell-free DNA fragmentation, copy number variations and the status of KRAS gene mutation, will be assessed to generate this model.

DETAILED DESCRIPTION:
The incidence of pancreatic cancer is insidious. Most patients were in advanced stage when diagnosed and could not be cured by surgery. Early diagnosis of pancreatic cancer through screening is so important. Early screening detection projects derived from liquid biopsy technology are not only limited to circulating DNA methylation markers, but have developed into multi-dimensional indicators for joint evaluation. This large-scale early detection study will randomly enroll 260 stage I/II/III pancreatic patients, 80 patients with pancreatic benign diseases and 156 age- and sex-matched healthy individuals upon providing written informed consent. Plasma samples will be collected and extracted cell-free DNA will be subjected to whole genome sequencing. We aimed to incorporate genome-wide copy number variations, cell-free DNA fragmentomics, and status of KRAS gene mutation into the development of a multimodal biomarker-based prediction model.

ELIGIBILITY:
Inclusion Criteria:

* Age minimum 18 years
* Participants must have histologically and/or cytologically confirmed stage I/II/III pancreatic cancer
* Full access to the patients' clinical and pathological records
* Ability to understand and the willingness to sign a written informed consent document
* Non-cancer controls are sex- and age-matched individuals without presence of any tumors or nodules or any other severe chronic diseases through systematic screening

Exclusion Criteria:

* Participants must not be pregnant or breastfeeding
* Participants must not have prior cancer histories or a second non-pancreatic malignancy
* Participants must not have had any form of cancer treatment before enrollment or plasma collection, including surgery, chemotherapy, radiotherapy, targeted therapy and immunotherapy
* Participants must not present medical conditions of fever or have acute or immunological diseases that required treatment 14 days before plasma collection
* Participants who underwent organ transplant or allogenic bone marrow or hematopoietic stem cell transplantation
* Participants with clinically important abnormalities or conditions unsuitable for blood collection
* Any uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, myocardial infarction, major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, or psychiatric illness/social situations that would limit compliance with study requirements or influence patient signing the written informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Approximately 260 stage I/II/III gastric cancer patients, 70 patients with pancreatic benign diseases and 150 non-cancer controls
Sampling Method: Non-Probability Sample
Enrollment: 496 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-10-12 (Estimated); Study Completion 2024-10-12 (Estimated)

PRIMARY OUTCOMES:
Area under curve of the model for detecting stage I/II/III pancreatic cancer | 2 years
  The area under curve of the model for the ultrasensitive early detection of stage I/II/III pancreatic cancer would be evaluate

SECONDARY OUTCOMES:
Sensitivity of the early detection modell | 2 years
  The sensitivity of the model for the ultrasensitive early detection of stage I/II/III pancreatic cancer would be evaluate
Specificity of the early detection model | 2 years
  The specificity of the model for the ultrasensitive early detection of stage I/II/III pancreatic cancer would be evaluate

CONTACTS AND LOCATIONS:
Overall Officials: Gao Chuntao, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No